CLINICAL TRIAL: NCT05972499
Title: Therapeutic Outcomes of Task-oriented Training With Pretend Play in Children With Cerebral Palsy.
Brief Title: the Effectiveness of Task-oriented Training With Pretend Play in CP Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, naira mohammed mosaad abdelmonem, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012004082
Record Dates: First submitted 2023-02-16; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (control group) (Placebo Comparator): The children in this group will receive physical therapy exercises to improve gross motor function and functional performance for 30 minutes per session ,3 times per week for three successive months as the following:
  Forward and sideways walking between parallel bars, as well as walking training with a stepper. Obstacles such as rolls and wedges are placed across the walking track during gait training in an open manner
  Interventions: Other: task-oriented training with pretend play
- Group B (study group) (Active Comparator): Task-oriented training with pretend play treatment:
  Individual interviews will be conducted with subjects and their parents to find their favorite story and to set up a pretend play situation for each subject. The child will have his specific script, will be constructed from his favorite story. The physical therapist will use modeling, prompts, and encouragement to initiate pretend play. Actions and verbalization on the scripts will be constructed to describe the performance of activities based on task-oriented training which include:
  Forward, sideways and backward walking. Walking through obstacle course. Walking up and down stairs. Walking up and down ramps. Running. Jumping. Each task will be given for 4 minutes and one minute rest. The child will be encouraged to complete the task and will be verbally cued during training. Tasks will be progressed according to each child's performance. These progressions included increasing the number of repetitions, and speed.
  Interventions: Other: task-oriented training with pretend play

INTERVENTIONS:
Other: task-oriented training with pretend play — Pretend play: Children engage in pretend play by acting out themes, taking on roles, assigning attributes to inanimate objects, and using objects as if they were something else Props will be added to hold the child interest. Role play costumes, or occupation props (police officer's suit), stimulate pretending elements.
  Task-oriented training: It is involving the active, repetitive practice of functional activities to learn or relearn a motor skill. Training implies that the behavioral experiences are not just repetition of the same sensorimotor skill but involves progressive challenges to a participant's capabilities and involves tasks that are meaningful to the participant. It is based on the following principles: functional goal-directed training focus on practicing specific activities of importance to the child during daily activities; planning activity-focused interventions by adapting knowledge of motor learning ; and allowing for the interest and participation of the children.

SUMMARY:
the effectiveness of task - oriented training with pretend play on gross motor function, functional capacity and cognitive function in children with hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
PURPOSE: This study aims to investigate the effectiveness of task-oriented training with pretend play on: gross motor function, functional capacity and cognitive function in children with hemiplegic CP.

BACKGROUND: Children with HCP experience difficulty with the motor function of the affected lower extremity. The majority of children with hemiplegia are able to walk without restrictions but more advanced gross motor skills are often affected.

Task-Oriented Training is a contemporary neurological rehabilitation technique that has the prospects of improving the quality of life of children with CP. It is a function-based, goal directed intervention that requires active involvement of the patient in a therapy that is task and context-specific, which focused on the accomplishment of functional activities and participation.

Pretend play is defined as play in which the child acts with intent that is representational. pretend play helps children learn how to express themselves, explore social interactions, and understand things and people within a real-world context.

HYPOTHESES: There is effect of task-oriented training with pretend play on gross motor function, functional capacity and cognitive function in children with hemiplegic CP.

. ………………… RESEARCH QUESTION: Does task-oriented training with pretend play has an effect on gross motor function, functional capacity and cognitive function in children with hemiplegic CP?

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic CP children of both genders.
* Their age range will be from 6 up to 8 years.
* They will be have spasticity will range from 1+ and 2, spasticity will be diagnosed based on the modified Ashworth scale.
* They will be have gross motor function at levels II and III, gross motor function will be diagnosed based on Gross Motor Function Classification System Expanded and Revised.
* They will be able to understand and follow direction.

Exclusion Criteria:

* Any visual or auditory impairments.
* Epilepsy.
* Any cognitive disorder.
* Any fracture or orthopedic surgery in the last 6 months.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
change from baseline in cognitive function on Wechsler intelligence scale for children (WISC-IV) at week13 | Baseline and week 13
  WISC-IV is a valid instrument assessing cognitive function. It consists of 10 core subtests and 5 supplementary subtests. it provides four index scores, The Full-Scale Intelligent Quotient can be obtained from the sum of the 10 core sub test scores.
  change= (Week 13 score - Baseline score).
change from baseline in functional capacity on six minutes walk test at week 13 | Baseline and week 13
  six minutes walk test is a validated instrument assessing functional capacity. For the 6 - minute walking test during overground walking, the children will be encouraged to walk on 30 meters hard and even surface corridor for 6- minutes .
  Change = (week 13 score -Baseline score).
change from baseline in gross motor function on Gross Motor Function Measure (GMFM) at week 13 | Baseline and week 13
  Gross Motor Function Measure is a valid, and reliable standardized assessment tool that measures change in gross motor function. It consists of 88 items grouped into five functional dimensions. Score of each item has four points ranging from 0 to 3; where 0 indicates that the child does not initiate the task; 3 indicates that the child completes the task (100%).
  change = (week 13 score -Baseline score).

IPD SHARING:
Plan to Share IPD: Undecided